CLINICAL TRIAL: NCT00647283
Title: ASSESSMENT OF THE SAFETY AND BENEFIT OF PROSPECTIVE IMMUNOSUPPRESSIVE DRUG WITHDRAWAL IN LIVER TRANSPLANTATION AND PREDICTION OF OPERATIONAL TOLERANCE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hospital Clinic of Barcelona (Other)
Collaborators: Fondo de Investigacion Sanitaria (Other); European Commission (Other); TcLand Expression S.A. (Industry)
Responsible Party: Alberto Sanchez-Fueyo, Hospital Clinic Barcelona / IDIBAPS
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: V-2005-CE512090-O; RISET
Record Dates: First submitted 2008-03-26; First posted 2008-03-31 (Estimated); Last update posted 2011-04-20 (Estimated); Status verified 2011-04

CONDITIONS: Liver Transplantation
Keywords: Liver Transplantation; Tolerance; Allograft tolerance; Immunosuppression minimization; Immunosuppression weaning; Immunological tolerance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Stable liver transplant recipients fulfilling inclusion criteria.
  Interventions: Procedure: Gradual immunosuppression drug withdrawal

INTERVENTIONS:
Procedure: Gradual immunosuppression drug withdrawal — After the obtention of biological samples (peripheral blood, liver tissue), enrolled patients undergo gradual weaning of all immunosuppressive therapy over a 6-9 month period under close medical supervision.

SUMMARY:
In liver transplantation up to 20% of recipients can completely discontinue immunosuppressive therapy maintaining normal graft function, and are conventionally considered as operationally tolerant. Discontinuation of immunosuppressive drugs in operationally tolerant recipients could lessen the side effects of chronic immunosuppressive therapy. However, this strategy results in the development of rejection in a high proportion of recipients who require lifelong immunosuppression. Thus, there is a need to identify predictive factors of successful drug withdrawal and to define the clinical and histological outcomes of operationally tolerant liver recipients.

The main objective of this study is to establish the safety of attempting immunosuppressive (IS) drug withdrawal in stable liver transplant recipients, using standard clinical, biological and histopathological methods, to screen and follow-up patients, and to confirm the benefit of maintaining immunosuppressive drug interruption in patients who are tolerant to their liver transplant. The secondary objective of this study is to identify predictive factors of operational tolerance and to attempt to develop a multi-parameter "decision rule" to predict patient tolerance or non-tolerance in order to improve patient screening and follow-up. In a diagnostic observational sub-study, peripheral blood and liver tissue samples collected before immunosuppressive drug withdrawal will be employed to validate the diagnostic accuracy of a previously identified set of tolerance biomarkers and to identify potential new biomarkers capable of predicting the outcome of the immunosuppressive withdrawal protocol.

DETAILED DESCRIPTION:
1. This is a prospective study in which liver transplant recipients on maintenance immunosuppression (IS) will undergo carefully supervised IS weaning over a period of approximately 6-9 months. Patients will be gathered from a consortium of European liver transplant units including: Hospital Clínic Barcelona (Dr A. Sánchez-Fueyo), University Tor Vergata Rome (Dr G.Tisone), University Hospitals Leuven (Dr J.Pirenne). Patients will be followed-up for a total of 48 months after inclusion.
2. Patients will be visited every 2-3 weeks, and immunosuppressive drugs will be gradually discontinued with the aim of achieving 50% decrease in drug dosages by month 3, and complete withdrawal by month 6 after initiation of the study. Following drug discontinuation, patients will continue to be followed every 2-3 weeks for 3 months, and monthly thereafter until month 12 after initiation of the study. Liver function tests will be obtained at every clinical follow-up visit. Patients will be considered operationally tolerant if no rejection takes place during the weaning procedure and the 12-month period after complete drug discontinuation. All patients who fail to completely discontinue IS, or in whom drugs have to be reintroduced after a period of complete withdrawal, are considered as IS-dependent or non-tolerant. All biopsies will be blindly reviewed at the end of the study by a single pathologist to ensure diagnostic consistency between the two institutions.
3. Management of liver function test alterations:

   * Increases in liver function tests below 2-fold normal levels for AST/ALT/GGT, 1.5-fold normal levels for ALP, or 2 mgIdL for bilirubin will result in no further decreases in drug dosages, and performance of new liver function tests in 14 days. Worsening or persistence of liver function test alterations will constitute indication for liver biopsy.
   * Increases in liver function tests beyond 2-fold normal levels for AST/ALT/GGT, 1.5-fold normal levels for ALP, or 2 mg/dL for bilirubin will result in liver biopsy.
4. Diagnosis of liver graft rejection: will be based on the finding of 2 out of 3 of the following histological criteria: portal inflammation, injury to bile duct epithelium, and endothelitis. The finding of a mixed portal/lobular lymphocytic infiltrate not attributable to any other cause and responding to an increase in immunosuppressive drug doses will also be considered as a rejection.
5. Management of rejection episodes: Specific therapy will be decided by the corresponding clinician/institution. Patients undergoing graft rejection will finalize their participation in the study. Worsening of HCV hepatitis or appearance of portal/lobular inflammation not attributable to rejection or viral etiology may also justify withdrawal from the study according to each institution's experience.
6. Peripheral blood samples will be collected before weaning starts and every time routine liver function tests are measured. These samples will be employed to conduct microarray gene expression experiments. A portion of all liver biopsies collected will also be cryopreserved to conduct gene expression analyses. This experiments will constitute the basis of an observational sub-study (described in a different protocol) entitled: "Search for the immunological signature of operational tolerance in liver transplantation".
7. Sample size has been estimated in order to be able to replicate the microarray gene expression results obtained by our group when comparing tolerant and non-tolerant recipients. In the current project we have followed a novel method recently proposed by Tibshirani et al. and have performed a permutation-based analysis of our pilot microarray data obtained from tolerant and non-tolerant samples. According to this analysis, at least 45 samples (20% tolerant, 80% non-tolerant) are required in order to be able to discriminate between tolerant and non-tolerant HCV-positive samples with a false discovery rate <0.05. Based on this analysis, we expect to enrol a total of 80 patients in order to have at least 60 patients evaluable, who will be randomly allocated into training (45 patients) and testing (15 patients) sets for data analysis purposes.

ELIGIBILITY:
Inclusion Criteria:

* Liver transplantation performed for non-autoimmune liver disease performed at least 3 years before IS weaning.
* Absence of acute and/or chronic rejection episodes during the 12 months before weaning.
* Basal liver biopsy without signs of acute and/or chronic rejection.
* No evidences of autoimmune liver disease.
* Absence of acute and/or chronic rejection episodes during the 12 months before weaning.
* Basal liver biopsy without signs of acute and/or chronic rejection.
* Low dose immunosuppression (monotherapy with calcineurin inhibitors, mTOR inhibitors or mycophenolate mofetil, or combined therapy with 2 drugs at very low doses).
* Absence of medical or psychological disturbances that preclude the safe performance of the trial.
* Stability of liver graft function, defined as: normal liver function tests (AST, ALT, ALP, GGT) during at least 6 months, or, alternatively, minor alterations in liver function tests that have not changed over the previous 6 months (AST/ALT < 2 fold normal levels; ALP < 1.5 fold normal levels; GGT < 2 fold normal levels; bilirubin < 2 mg/dL).
* Patients exhibiting at least one of the following characteristics: a) severe side effects of immunosuppressive drugs (diabetes, renal failure, hyperlipidemia, hypertension); b) risk of neoplasm development defined by history of previous non-hepatocarcinoma neoplasms or history of any of the following risk factors: tobacco or alcohol consumption, age greater than 60 years; c) chronic liver disease due to hepatitis C virus infection in patients not receiving anti-viral treatment.
* Signature of informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2005-11; Primary Completion 2010-09 (Actual); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Operational tolerance defined as liver transplant survival with immunosuppressive drug interruption and without liver transplant rejection after starting drug dose reduction and following 12 months of complete drug discontinuation. | 18 months

SECONDARY OUTCOMES:
Prevalence of patients developing permanent graft dysfunction as a consequence of immunosuppressive drug withdrawal. | 48 months
Effects of the immunosuppression weaning procedure on immunosuppression-related side effects (hypertension, diabetes, nephrotoxicity, hyperlipidemia) | 48 months

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Sanchez-Fueyo, MD, Principal Investigator — Hospital Clinic Barcelona / IDIBAPS, Barcelona, Spain; Giuseppe Tisone, MD, Study Chair — University Tor Vergata, Rome, Italy; Jacques Pirenne, MD, Study Chair — Abdominal Transplant Surgery Department, University Hospitals Leuven, Belgium
Locations (1):
- Hospital Clinic Barcelona, University of Barcelona, Barcelona, Barcelona, Spain

REFERENCES:
- [Background] Martinez-Llordella M, Puig-Pey I, Orlando G, Ramoni M, Tisone G, Rimola A, Lerut J, Latinne D, Margarit C, Bilbao I, Brouard S, Hernandez-Fuentes M, Soulillou JP, Sanchez-Fueyo A. Multiparameter immune profiling of operational tolerance in liver transplantation. Am J Transplant. 2007 Feb;7(2):309-19. doi: 10.1111/j.1600-6143.2006.01621.x. PMID 17241111